CLINICAL TRIAL: NCT05615870
Title: Bronchiolitis Recovery and the Use of High Efficiency Particulate Air (HEPA) Filters
Acronym: BREATHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IDeA States Pediatric Clinical Trials Network (Network)
Collaborators: University of Vermont Medical Center (Other); University of Montana (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 274137; U24OD024957 (NIH)
Record Dates: First submitted 2022-09-17; First posted 2022-11-14 (Actual); Results first posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Bronchiolitis
Keywords: Children<12 months of age hospitalized with bronchiolitis
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Intervention Model Description: This is a multi-center, parallel, double-blind, randomized controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Families will be masked as to whether their Winix units are equipped with or without HEPA/carbon filters.
  Study coordinators, investigators, and other team members who interact with participants' parent(s)/guardian(s) to obtain surveys, troubleshoot equipment setup and operation, or have other interactions will remain masked through the duration of the study for individual participants. This includes masking as to which intervention the participants receive and household air quality measurements, including the baseline measurements (separate personnel will need to be on the receiving end for air quality measurement data). This will require more than one study coordinator or additional staff/technician on the study team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Filter) (Active Comparator): The intervention group will use two Winix 5500-2 HEPA filtration units (Appendix A) (https://winixamerica.com/product/5500-2/). One will be placed in the child's sleep space and one will be placed in another common room with both units running continuously on the "high" (i.e., level 3 / second from highest) setting. Each unit is 8.2 x 15.0 x 23.6 inches, and verified for a 360 sq. foot room. If a home is too small to accommodate 2 Winix units (for example, a single room residence'), one Winix unit may be used for the study. Additional features beyond HEPA and carbon filter, include plasmawave technology to reduce volatile organic compounds and odors. The plasmawave feature will be turned off to avoid ozone production.
  Interventions: Other: Winix 5500-2 HEPA filtration units
- Control Group (No Filter) (Sham Comparator): The control group will use identical-appearing Winix 5500-2 units and identical setup procedures as described above, but with no HEPA or carbon filters.
  Interventions: Other: Winix 5500-2 HEPA filtration units

INTERVENTIONS:
Other: Winix 5500-2 HEPA filtration units — To determine if use of a HEPA filtration unit home intervention reduces the respiratory symptom burden (symptom-free days; SFD) for 24 weeks compared to a use of a control unit.

SUMMARY:
This is a multi-center, parallel, double-blind, randomized controlled clinical trial. Children <12 months of age hospitalized with bronchiolitis are randomized 1:1 to receive a 24-week home intervention with filtration units containing HEPA and carbon filters (in the child's sleep space and a common room) to improve indoor air quality (IAQ) or to a control group with filtration units without HEPA and carbon filters. The HEPA intervention units and control units will be used for 24 weeks after pre-intervention IAQ measurements. Children are followed for respiratory outcomes over the pre-intervention and intervention periods.

DETAILED DESCRIPTION:
This is a multi-center, parallel, double-blind, randomized controlled clinical trial. Two hundred twenty-eight children <12 months old with their first hospitalization for bronchiolitis will be randomized 1:1 (stratified by site) to receive 24 weeks of home intervention with active HEPA filtration units to improve IAQ or to a control group without a HEPA or carbon filter inside identical-appearing units. Children will be followed for respiratory symptoms during a pre-intervention period of up to two weeks following randomization and during an intervention period of 24 weeks.

This study is designed to reduce barriers to participation for rural participants in that there will be no required study visits to a distant study site, and all study activities and data collection will be conducted remotely. Participants will be identified in hospitals in ISPCTN states, maximizing the chances that rural and medically underserved populations are represented. It is common for rural children with bronchiolitis to be transferred to tertiary care centers in urban/suburban locales, so inclusion of urban hospitals will allow for recruitment of this population.1 It is important for rural children to be represented in a bronchiolitis study in order to increase generalizability. Rural and underserved children have a higher risk of decreased access to medical care for symptoms and illness episodes, and a higher burden of asthma.83,84 These families may have air pollutant exposure profiles distinct from those residing in urban areas. For example, they might experience less exposure to traffic-related pollutants but may have more wood stove use or exposure to agricultural pollutants or wildfires. With its diversity of sites, the ECHO ISPCTN is well-positioned to enroll rural children that might otherwise be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Age <12 months at hospital admission
* First-time hospitalization for bronchiolitis
* One primary residence (>5 days per week)
* Parent, legal guardian or other legally authorized representative consents to allow their child to participate and agrees to participate in all study activities
* Electricity in the home (required to power the study equipment)
* Wireless internet access or cellular service access in the home*
* English or Spanish-speaking parent or guardian

Exclusion Criteria:

* Chronic airway or respiratory conditions requiring home oxygen, mechanical ventilation, or tracheostomy dependence; known immunodeficiency, hemodynamically significant cardiac conditions including those requiring medication or oxygen; cystic fibrosis; neuromuscular disease; eligible for palivizumab (per AAP guidelines87)
* Use of stand-alone home HEPA filtration other than study-related HEPA units in the home
* Household member who smokes (any type), vapes, or uses e-cigarettes
* Intention to move in the next 6 months
* Enrolled or plans to enroll in an interventional clinical trial for treatment of acute bronchiolitis or sequelae of bronchiolitis, unless permission given by the PI
* Another child in the household is enrolled in this study (one child per household can enroll)

Ages: 1 Week to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 230 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Cowan, MD, Study Chair — University of Vermont Medical Center; Erin Semmens, PhD, MPH, Study Chair — University of Montana
Locations (17):
- United States (17):
  - Alaska Native Tribal Health Consortium, Anchorage, Alaska
  - Arkansas Children's Hospital - Little Rock (ACHRI), Little Rock, Arkansas
  - Kapi'olani Medical Center for Women and Children, Honolulu, Hawaii
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Tulane University, Department of Pediatrics, New Orleans, Louisiana
  - University of Miss. Medical Center, Jackson, Mississippi
  - University of Montana, Missoula, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hospital, Lebanon, New Hampshire
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - Children's Hospital OU Medical Center, Oklahoma City, Oklahoma
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health-Midlands, Columbia, South Carolina
  - Avera Research Institute, Sioux Falls, South Dakota
  - University of Vermont Medical Center, Burlington, Vermont
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
The study team will place participant's de-identified data and other limited information, such as race and ethnic group, into one or more centralized database(s). The study team will share this data in compliance with the ISPCTN and NIH data sharing policies
Supporting Information: SAP
Time Frame: NIH Public Access Policy ensures public access to the published results of NIH-funded research. Scientists are required to submit final peer-reviewed journal manuscripts from NIH funds to the digital archive PubMed Central upon publication acceptance.
  ECHO ISPCTN Publications and Presentations Policy, ensures accurate, responsible, and efficient communication of findings from ECHO ISPCTN clinical trials. The ECHO ISPCTN Steering Committee has approved and ratified the Publications and Presentations Policy, which includes representatives from all site awardees, as well as representatives from NIH and the DCOC NIH Data Sharing Policy, the policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission Rule. Trial results will be submitted to ClinicalTrials.gov. Additional plans are to publish results in peer reviewed journals. Researchers may request trial data by contacting Jeannette Lee, PhD, at the DCOC.
Access Criteria: TBA

REFERENCES:
- [Derived] Cowan K, Semmens EO, Lee JY, Walker ES, Smith PG, Fu L, Singleton R, Cox SM, Faiella J, Chassereau L, Lawrence L, Ying J, Baldner J, Garza M, Annett R, Chervinskiy SK, Snowden J. Bronchiolitis recovery and the use of High Efficiency Particulate Air (HEPA) Filters (The BREATHE Study): study protocol for a multi-center, parallel, double-blind, randomized controlled clinical trial. Trials. 2024 Mar 20;25(1):197. doi: 10.1186/s13063-024-08012-0. PMID 38504367

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two enrolled participants terminated the study prior to randomization due to withdrawal of consent and ineligibility.
Period: Overall Study
Arm/Group | Intervention Group (Active Filter) | Control Group (No Filter)
Started | 113 | 115
Completed | 100 | 94
Not Completed | 13 | 21
Not completed — Lost to Follow-up | 10 | 13
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Protocol Violation | 0 | 3
Not completed — Unable to complete study activities after moving residences | 0 | 2
Not completed — Terminated from the experimental or control intervention only and continued with the study | 1 | 0
Not completed — The participant thought the study was done and shipped the devices back. | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all participants who are randomized to either the HEPA filtration (intervention group) or the inactive filter unit (control group).
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group (Active Filter) | Control Group (No Filter) | Total
Number analyzed (Participants) | 113 | 115 | 228
Age, Continuous [Mean (Standard Deviation); unit: Months] | 4.0 (2.9) | 4.3 (2.9) | 4.1 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 49 | 90
  Male | 72 | 66 | 138
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 12 | 28
  Not Hispanic or Latino | 94 | 102 | 196
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10 | 6 | 16
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 13 | 16 | 29
  White | 70 | 74 | 144
  More than one race | 16 | 14 | 30
  Unknown or Not Reported | 3 | 3 | 6
Rurality (RUCA code) [Count of Participants; unit: Participants] — Metropolitan: RUCA code<4 Micropolitan: 4<=RUCA cod<7 Small town: 7<=RUCA code<10 Rural area: RUCA code>=10
  Participants
    Metropolitan | 79 | 78 | 157
    Micropolitan | 9 | 14 | 23
    Small town | 5 | 12 | 17
    Rural | 19 | 9 | 28
    Unknown | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Caregiver-reported Symptom-free Days (SFDs)
Description: An SFD is defined as a 24-hour period without coughing, wheezing, or trouble breathing
Time Frame: 24 Weeks
Population: The analysis population included all participants who were randomized to either HEPA filtration (intervention group) or inactive filter unit (control group) with available outcome data
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Intervention Group (Active Filter) | Control Group (No Filter)
Number analyzed (Participants) | 110 | 109
Days | 118.01 (42.66) | 112.60 (46.33)
Statistical Analysis 1: Comparison: Intervention Group (Active Filter) vs Control Group (No Filter); Null hypothesis: mean of SFDs in the HEPA filtration home intervention group will not differ from the mean of SFDs in the control group; Test type: Superiority; p = 0.537, Mixed Models Analysis; Mean Difference (Final Values) = 5.41, 95% CI 2-sided [-11.77 to 22.60]

2. Secondary Outcome: Number of Hospitalizations, Emergency Department or Urgent Care Visits or Other Unscheduled Medical Visits for Respiratory Complaints
Description: Caregiver reported number of hospitalizations, emergency department or urgent care visits, other unscheduled medical visits, and the sum of total counts of all metrics for respiratory complaints
Time Frame: 24 weeks
Population: The analysis population included all participants who are randomized to either HEPA filtration (intervention group) or inactive filter unit (control group) with available data of Unscheduled Healthcare Visits
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | Intervention Group (Active Filter) | Control Group (No Filter)
Number analyzed (Participants) | 109 | 109
Visits
  Hospitalizations | 0.28 (0.91) | 0.16 (0.60)
  Emergency Department (ED) or Urgent Care (UC) visits | 0.68 (1.25) | 0.68 (1.32)
  Other unscheduled healthcare visits (UHVs) for respiratory complaints | 1.11 (1.65) | 1.48 (1.99)
  A sum of counts (or total counts) of all metrics | 2.06 (2.83) | 2.31 (2.84)
Statistical Analysis 1: Comparison: Intervention Group (Active Filter) vs Control Group (No Filter); Null hypothesis: mean of counts of hospitalizations for respiratory symptoms in the intervention group will not differ from the mean of counts of hospitalizations for respiratory symptoms in the control group; Test type: Superiority; p = 0.205, Mixed Models Analysis; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.07 to 0.30]
Statistical Analysis 2: Comparison: Intervention Group (Active Filter) vs Control Group (No Filter); Null hypothesis: mean of counts of emergency department or urgent care visits for respiratory symptoms in the intervention group will not differ from the mean of counts of emergency department or urgent care visits for respiratory symptoms in the control group; Test type: Superiority; p = 0.992, Mixed Models Analysis; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.35 to 0.35]
Statistical Analysis 3: Comparison: Intervention Group (Active Filter) vs Control Group (No Filter); Null hypothesis: mean of counts of other unscheduled healthcare visits for respiratory symptoms in the intervention group will not differ from the mean of counts of other unscheduled healthcare visits for respiratory symptoms in the control group; Test type: Superiority; p = 0.172, Mixed Models Analysis; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.90 to 0.16]
Statistical Analysis 4: Comparison: Intervention Group (Active Filter) vs Control Group (No Filter); Null hypothesis: mean of counts (or total counts) of visits of all metrics for respiratory symptoms in the intervention group will not differ from the mean of counts of visits of all metrics for respiratory symptoms in the control group; Test type: Superiority; p = 0.530, Mixed Models Analysis; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-1.02 to 0.52]

3. Secondary Outcome: Total Quality of Life (QOL) Score
Description: QOL score is measured by the Pediatric Quality of Life Inventory TM (PedsQLTM) Infants Scales questionnaire. The scores are reverse-scored and linearly transformed to a 0-100 scale. Higher scores mean a better outcome.
Time Frame: 24 weeks
Population: Participants who were randomized to either HEPA filtration (intervention group) or inactive filter unit (control group) and answered the quality of life (QOL) survey.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Intervention Group (Active Filter) | Control Group (No Filter)
Number analyzed (Participants) | 100 | 95
Scores on a scale | 81.34 (9.99) | 82.13 (10.68)
Statistical Analysis 1: Comparison: Intervention Group (Active Filter) vs Control Group (No Filter); Null hypothesis: mean of the Child QOL score in the HEPA intervention group will not differ from the mean of Child QOL score in the control group; Test type: Superiority; p = 0.598, Mixed Models Analysis; Mean Difference (Final Values) = -0.80, 95% CI 2-sided [-3.75 to 2.16]

4. Secondary Outcome: Average Particulate Matter (PM2.5) Levels
Description: PM2.5 levels (Particulate Matter ≤ 2.5 micrometers in diameter) are measured by in-home monitors and scaled to unit of micrograms per cubic meter per week. Higher levels mean a worse outcome.
Time Frame: 24 weeks
Population: Participants who were randomized to either HEPA filtration (intervention group) or inactive filter unit (control group) with available PM2.5 data
Measure: Mean (Standard Deviation); unit: µg/m³/week
Arm/Group | Intervention Group (Active Filter) | Control Group (No Filter)
Number analyzed (Participants) | 102 | 100
µg/m³/week
  Common room: number analyzed (Participants) | 98 | 96
  Common room | 10.70 (15.91) | 15.27 (16.86)
  Sleep space: number analyzed (Participants) | 95 | 96
  Sleep space | 11.08 (18.77) | 21.45 (33.14)
  Average of common room and sleep space | 10.66 (15.53) | 17.96 (21.35)
Statistical Analysis 1: Comparison: Intervention Group (Active Filter) vs Control Group (No Filter); Null hypothesis: the mean of the PM2.5 level of the common room and sleep space in the intervention group will not differ from the mean of the PM2.5 level in the control group; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -7.20, 95% CI 2-sided [-10.98 to -3.42] — The results were based on the average PM2.5 level of common room and sleep space

ADVERSE EVENTS:
Time Frame: From November 24, 2022, to May 22, 2024 (1 year, 5.9 months)
Arm/Group | Intervention Group (Active Filter) | Control Group (No Filter)
All-Cause Mortality (participants affected / at risk) | 0/113 | 0/115
Serious Adverse Events (participants affected / at risk) | 17/113 | 12/115
Other Adverse Events (participants affected / at risk) | 7/113 | 11/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Group (Active Filter) (N=113) | Control Group (No Filter) (N=115)
Medical or emergency department/urgent care visit for respiratory complaint (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Trouble breathing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Wheeze (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Other - bronchiolitis, hospitalization for hypoxia & increased work of breathing, and respiratory di (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Other - Respiratory Distress, Reactive airway disease with wheezing, Hypoxemia and nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Other - Bronchiolitis (Infections and infestations) | 6 | 5
Other - seizure like activity (Nervous system disorders) | 1 | 0
VSD repair surgery (Surgical and medical procedures) | 1 | 0
Other - Patient had bilateral ear tubes placed (Injury, poisoning and procedural complications) | 1 | 0
Other - Hospitalization due to failure to thrive (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Group (Active Filter) (N=113) | Control Group (No Filter) (N=115)
Other - Subglottic stenosis requiring micro laryngoscopy and bronchoscopy / Reactive Airway Disease (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Medical or emergency department/urgent care visit for respiratory complaint (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Other - Rhinitis, Coughing, Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Other - Cough (Infections and infestations) | 1 | 1
Other- Viral induced asthma (Immune system disorders) | 0 | 2
Other - Constipation issues that required emergency room visit (Gastrointestinal disorders) | 0 | 1
Other - Seizure (Nervous system disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-09-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT05615870/Prot_002.pdf
  • Statistical Analysis Plan (2025-04-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT05615870/SAP_003.pdf
  • Informed Consent Form (2023-08-30): https://cdn.clinicaltrials.gov/large-docs/70/NCT05615870/ICF_001.pdf